CLINICAL TRIAL: NCT05623618
Title: A Cluster Randomised Controlled Trial Testing Physical Activity Calorie Equivalent (PACE) Labelling on Discretionary Foods in Secondary Schools
Brief Title: Understanding the Impact of Physical Activity Calorie Equivalent (PACE) Labelling in Secondary Schools
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Loughborough University (Other)
Collaborators: Natalia Iris (Unknown)
Responsible Party: Principal Investigator, Amanda Daley, Professor, Loughborough University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 7011
Record Dates: First submitted 2022-10-13; First posted 2022-11-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Eating Behaviour of Discretionary Foods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (PACE labelling) (Experimental): PACE labelling implemented near at least one discretionary food item in secondary school canteens for up to 6 weeks.
  Interventions: Behavioral: PACE labelling
- Control (usual practice) (No Intervention): PACE labelling not implemented. Secondary schools continue with their usual practice.

INTERVENTIONS:
Behavioral: PACE labelling — PACE labelling implemented near at least one discretionary food item in secondary school canteens for up to 6 weeks.
  Arms: Intervention (PACE labelling)

SUMMARY:
The aim is to undertake a cluster randomised controlled trial to assess the effectiveness of PACE food labelling in reducing young people's purchasing of discretionary foods in secondary school canteens. Physical activity calorie equivalent (PACE) food labelling aims to show the number of minutes or miles/kilometres of physical activity equivalent to the calories contained in food/drinks.

DETAILED DESCRIPTION:
Physical activity calorie equivalent (PACE) food labelling aims to show the number of minutes or miles/kilometres of physical activity equivalent to the calories contained in food/drinks. Evidence suggests that PACE food labelling may influence food/drink choice. Most research in this area however have tested PACE food labels with adults and/or have tested hypothetical food choice scenarios. Studies in real world contexts with young people are needed to see if PACE food labels could help them make healthier food choices.

The aim is to assess the effectiveness of PACE food labelling in reducing young people's purchasing of discretionary foods in secondary school canteens. A cluster randomised controlled trial with a nested qualitative study will be conducted. Secondary schools will be randomised to either display PACE labelling near discretionary foods or continue with their usual practice. The intervention period will be up to 6 weeks. Anonymised purchase data will be collected throughout the study period.

Qualitative interviews will be conducted with students in the intervention schools to explore their views of the PACE labels such as perceived influence of the PACE labelling on their food selection.

ELIGIBILITY:
Secondary schools:

Inclusion Criteria:

* Secondary schools that admit young people aged between 10 to 19 years.
* Sell at least one type of cake and/or at least one type of sweet biscuit for at least 2 days per week up to a 6 week period (or equivalent), and have sold the same cake(s)/biscuit(s) before the study (for a minimum of 4 weeks).
* Able to provide to the researcher with anonymised purchase data for study periods. Data to include number of units sold and dates sold of the chosen food item(s).
* A PACE label could feasibly be placed near to the study elected food item(s) in a school canteen used by students.
* Not participating in any other school trials or initiatives.

Exclusion Criteria:

* Secondary schools not meeting the inclusion criteria.
* Secondary schools that admit young people below the age of 10 years or above the age of 19 years.

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 8000 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Change in number of daily purchases/units sold of the specified discretionary food(s) in secondary school canteens. | Baseline period (a minimum of 4 weeks), Intervention period (up to 6 weeks) and Washout period (up to 6 weeks, and if time allows)

CONTACTS AND LOCATIONS:
Locations (1):
- Loughborough University, Loughborough, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iris N, Munir F, Daley AJ. Physical activity calorie equivalent (PACE) food labelling on discretionary foods in secondary school canteens in England: an efficacy cluster randomised controlled trial. Int J Behav Nutr Phys Act. 2025 Feb 26;22(1):24. doi: 10.1186/s12966-025-01710-1. PMID 40011948